CLINICAL TRIAL: NCT00006486
Title: A Phase II Randomized Discontinuation Trial Of Carboxyaminoimidazole (CAI, NSC 609974) In Metastatic Renal Carcinoma
Brief Title: Carboxyamidotriazole in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02364; CLB-69901; U10CA031946 (NIH); CDR0000068317 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-11-06; First posted 2003-07-28 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — carboxyamido-triazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (carboxyaminoimidazole) (Experimental): Patients receive oral CAI daily for 4 weeks. Treatment repeats for 4 courses in the absence of disease progression or unacceptable toxicity. After 4 courses, patients experiencing complete or partial response continue treatment until disease progression or unacceptable toxicity.
  Patients receive oral CAI as above.
  Interventions: Drug: carboxyamidotriazole
- Arm II (carboxyamidotriazole, placebo) (Experimental): Patients receive oral CAI daily for 4 weeks. Treatment repeats for 4 courses in the absence of disease progression or unacceptable toxicity. After 4 courses, patients experiencing complete or partial response continue treatment until disease progression or unacceptable toxicity.
  Patients receive a placebo.
  Interventions: Drug: carboxyamidotriazole; Other: placebo

INTERVENTIONS:
Drug: carboxyamidotriazole — Given orally
  Other Names: CAI; carboxyamido-triazole; carboxyaminoimidazole
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (carboxyamidotriazole, placebo)

SUMMARY:
Randomized phase II trial to study the effectiveness of carboxyamidotriazole in treating patients who have metastatic kidney cancer. Carboxyamidotriazole may stop the growth of kidney cancer by stopping blood flow to the tumor

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxicity and disease-stabilizing effect of carboxyamidotriazole in patients with metastatic renal cell carcinoma.

II. Determine the objective response rate in patients treated with this drug.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to time from diagnosis of metastatic disease to study entry (fewer than 24 months vs 24 months or more).

Patients receive oral carboxyamidotriazole (CAI) daily for 4 weeks. Treatment repeats for 4 courses in the absence of disease progression or unacceptable toxicity. After 4 courses, patients experiencing complete or partial response continue treatment until disease progression or unacceptable toxicity.

Patients with stable disease are randomized to one of two treatment arms.

Arm I: Patients receive oral CAI as above.

Arm II: Patients receive a placebo.

Treatment repeats every 4 weeks for at least 4 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression are unblinded and those on placebo begin oral CAI as above.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A maximum of 335 patients will be accrued for this study within 15-25 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma

  * Metastatic or unresectable disease
  * Documented disease progression, even after nephrectomy
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * The following lesions are not considered measurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses not confirmed and followed by imaging
    * Cystic lesions
* Performance status - CTC 0-2
* WBC at least 2,000/mm^3
* Platelet count at least 75,000/mm^3
* Bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Creatinine no greater than 2.0 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No baseline neuropathy or cerebellar dysfunction greater than grade 1
* At least 4 weeks since prior immunotherapy
* No prior carboxyamidotriazole
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* Concurrent epoetin alfa allowed
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy
* No concurrent hormonal therapy except steroids for adrenal failure or hormones for conditions not related to disease (e.g., insulin for diabetes)
* At least 4 weeks since prior radiotherapy
* No concurrent palliative radiotherapy
* See Disease Characteristics
* At least 4 weeks since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2000-10; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients progressing on placebo to the proportion progressing on CAI | Up to 16 weeks
Proportions of patients with stable disease | Up to 16 weeks
Objective response | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States